CLINICAL TRIAL: NCT06937307
Title: Droxidopa to Increase Mean Arterial Pressure in Decompensated Cirrhosis Patients With Acute Kidney Injury
Acronym: DROP-AKI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Giuseppe Cullaro, MD (Other)
Responsible Party: Sponsor-Investigator, Giuseppe Cullaro, MD, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAV7484
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Acute Kidney Injury; Cirrhosis; Decompensated Cirrhosis of Liver
Keywords: Acute Kidney Injury; Cirrhosis; Decompensated Cirrhosis
MeSH Terms: conditions — Acute Kidney Injury; Fibrosis | interventions — Droxidopa; 3,4-dihydroxyphenylserine aldolase

STUDY DESIGN:
Intervention Model Description: This study employs a parallel-group design where hospitalized patients with decompensated cirrhosis and acute kidney injury are randomized in a 2:1 ratio to receive either droxidopa or matching placebo. Both groups will receive the intervention concurrently over the 28-day treatment period, with identical titration protocols and assessment schedules. Participants in the active arm will receive droxidopa initially at 100 mg three times daily, titrated based on mean arterial pressure response, while the control arm will receive identical-appearing placebo capsules following the same schedule and titration protocol to maintain blinding.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind, placebo-controlled study in which both active drug (droxidopa) and placebo will be over-encapsulated using identical opaque capsules by the Columbia University Research Pharmacy. Only the Research Pharmacy staff will be unblinded to enable proper preparation and dispensing of study medication, while all participants, investigators, care providers, and outcomes assessors will remain blinded to treatment assignment. Emergency unblinding procedures are available through the Research Pharmacy if needed for subject safety, but otherwise the blind will be maintained until study completion and database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Droxidopa (Experimental): Participants in this arm will receive oral droxidopa capsules at an initial dose of 100 mg three times daily, titrated in 100 mg increments every 24 hours based on blood pressure response and tolerability, up to a maximum dose of 300 mg three times daily. Doses will be given approximately 4 hours apart during daytime hours for a total treatment duration of 28 days.
  Interventions: Drug: Droxidopa capsules
- Placebo (Placebo Comparator): Participants in this arm will receive matched placebo capsules following the same dosing schedule and titration protocol as the experimental arm. Placebo capsules will be identical in appearance to droxidopa capsules with the same over-encapsulation process to maintain blinding. Doses will be given three times daily for a total treatment duration of 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Droxidopa capsules — Droxidopa is an oral synthetic amino acid that is directly metabolized to norepinephrine by dopa-decarboxylase. It will be administered at an initial dose of 100 mg three times daily, titrated in 100 mg increments every 24 hours based on blood pressure response, up to a maximum of 300 mg three times daily. Doses will be given approximately 4 hours apart during daytime hours, at least 3 hours apart, with a maximum total daily dose of 900 mg. The treatment duration is 28 days. The drug will be over-encapsulated using opaque capsules to maintain the double-blind design.
  Other Names: L-threo-3,4-dihydroxyphenylserine
  Arms: Droxidopa
Other: Placebo — Matching placebo capsules containing microcrystalline cellulose (from Millipore Sigma) will be over-encapsulated using identical opaque capsules to maintain blinding. Placebo will be administered following the same schedule as the active treatment: three times daily with the same titration protocol based on blood pressure response, for a treatment duration of 28 days. The Columbia University Research Pharmacy will perform over-encapsulation of both active drug and placebo to ensure they are identical in appearance.
  Arms: Placebo

SUMMARY:
This study tests whether a medication called droxidopa can help improve blood flow to the kidneys in people with liver cirrhosis who develop kidney problems while in the hospital. When someone with cirrhosis experiences kidney injury, having better blood pressure can help their kidneys recover. Droxidopa is an oral medication that may help raise blood pressure without requiring intensive care or invasive treatments. The study will compare droxidopa to a placebo (inactive pill) in 75 people hospitalized with cirrhosis and kidney injury. Participants will take either droxidopa or placebo pills for 28 days and be monitored for an additional 30 days. Researchers will measure changes in blood pressure and kidney function to determine if droxidopa is effective and safe for these patients. This research could identify a new treatment option for a serious complication of liver disease.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) occurs in up to 50% of hospitalized patients with decompensated cirrhosis and carries mortality rates exceeding 50%. Recent evidence indicates that progression of AKI after initial diagnosis significantly impacts outcomes, with patients whose AKI worsens having up to 8 times higher mortality compared to those without progression.

Mean arterial pressure (MAP) appears to be a key mediator of kidney function and recovery in cirrhosis. Multiple studies have established that each 5 mmHg increase in MAP is associated with a 1.07-1.19 times greater likelihood of AKI recovery. However, current therapeutic options to increase MAP in cirrhosis are limited to invasive vasopressors requiring ICU admission, terlipressin with significant risks including respiratory failure, or oral midodrine which lacks proven efficacy in decompensated cirrhosis.

Droxidopa is an oral synthetic amino acid that is directly metabolized to norepinephrine by dopa-decarboxylase. FDA-approved since 2014 for neurogenic orthostatic hypotension, droxidopa demonstrates a well-established safety profile and consistent ability to increase systolic blood pressure by 7-11 mmHg. This magnitude of effect is similar to that associated with AKI recovery when using invasive vasopressors. Importantly, droxidopa maintains efficacy over 12 weeks with minimal risk of supine hypertension.

This study will evaluate droxidopa in a 2:1 randomized, double-blind, placebo-controlled trial of 75 hospitalized patients with Child-Pugh Score ≥B7 cirrhosis and KDIGO Stage 1 AKI or greater who have MAP ≤85 mmHg. Participants will receive droxidopa or placebo initially at 100 mg three times daily, titrated in 100 mg increments every 24 hours based on blood pressure response and tolerability, up to a maximum of 300 mg three times daily for 28 days.

The primary endpoint is change in MAP, measured by a linear mixed-effects model with fixed effects for treatment group and time. Secondary endpoints include change in serum creatinine, completion of study day 28, death, and liver transplantation. Safety will be carefully monitored with primary safety endpoints of hypertensive emergency and development of cardiac arrhythmias.

An Internal Data and Safety Monitoring Board consisting of an independent hepatologist with cirrhosis expertise, a biostatistician experienced in clinical trials, and a study medical monitor will review safety data monthly and assess stopping rules criteria.

Total study duration will be 58 days (28 days of product administration plus 30 days of follow-up) per participant, with an overall study timeline of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent by subject or legally authorized representative
* Consent to blood and urine collection for biomarker analysis
* Ability to take oral medications
* At least 18 years of age
* Hospitalized at Columbia University Irving Medical Center
* Child-Pugh Score ≥ B7 cirrhosis (documented by imaging, biopsy, or clinical evidence)
* KDIGO Stage 1 AKI or greater, defined as:
* ≥0.3 mg/dL increase in serum creatinine within 48 hours OR
* ≥50% increase in serum creatinine from outpatient baseline
* Mean arterial pressure ≤85 mmHg averaged over 24 hours prior to randomization
* For women of childbearing potential: negative pregnancy test and agreement to use effective contraception

Exclusion Criteria:

* Serum creatinine >4.0 mg/dL or current renal replacement therapy
* Age >70 years
* Severe cardiovascular disease, including:
* Unstable angina
* Congestive heart failure requiring escalating medical therapy
* Symptomatic peripheral vascular disease
* Any cardiovascular condition deemed severe by investigator
* Active gastrointestinal bleeding, defined as requiring ≥ 2 units of packed red blood cells during the screening period
* Acute respiratory failure requiring more than 6L of Nasal Canula
* Use of medications that could interact with droxidopa including:
* MAOI inhibitors
* Norepinephrine reuptake inhibitors
* Other investigational drugs
* Pregnancy or breastfeeding
* Any episode of a SBP ≥ 180 mmHg or a DBP ≥ 120 mmHg on two measurements, 1 minute apart
* Prior liver transplantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in mean arterial pressure (MAP) | Baseline to 28 days
  The difference in mean arterial pressure between treatment groups over the 28-day treatment period, assessed using a linear mixed-effects model with fixed effects for treatment group and time, plus their interaction, while accounting for between-subject variability through random intercepts.

SECONDARY OUTCOMES:
Change in serum creatinine | 28 days
  The difference in serum creatinine between treatment groups over the 28-day treatment period, assessed using a linear mixed-effects model with fixed effects for treatment group and time, plus their interaction, while accounting for between-subject variability through random intercepts.
All-cause mortality | 58 days
  The proportion of participants who die from any cause during the study period.
Liver transplantation | 58 days
  The proportion of participants who undergo liver transplantation during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Cullaro, MD, MAS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing decisions remain under institutional review. Key considerations include: (1) protecting sensitive health information for vulnerable cirrhosis patients, (2) aligning with Columbia University's data governance frameworks, (3) determining appropriate de-identification methodologies, and (4) developing suitable data dictionaries and transfer protocols. Upon study completion, a comprehensive data sharing determination will be made, with potential for de-identified datasets to be shared through secure repositories following primary publication.